CLINICAL TRIAL: NCT02809001
Title: The Effects of Autologous Fat Transfer on Preventing Expanded Skin From Expansion Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, Director of plastic and reconstructive surgery department, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Shanghai9PH
Record Dates: First submitted 2016-06-05; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Scar; Nevus
Keywords: Fat grafting; Expansion-related complications
MeSH Terms: conditions — Cicatrix; Nevus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Experimental: Fat grafting (Experimental): Autologous fat graft transplantation subdermally to expanded skin.
  Interventions: Procedure: Fat grafting
- Control (No Intervention): Expansion was discontinued until the early signs of complication disappeared.

INTERVENTIONS:
Procedure: Fat grafting — In the experimental group, liposuction will be performed and autologous fat graft will be harvest after washing with saline. Patients will receive autologous fat graft transplantation subdermally to expanded skin.
  Arms: Experimental: Fat grafting

SUMMARY:
The purpose of this study is to evaluate whether autologous fat grafting is safe and/or effective to prevent expanded skin from expansion failure.

DETAILED DESCRIPTION:
The repair of skin defects is a common problem for reconstructive surgeons.Soft tissue expansion is a widely used technique for the repair of skin defects. Early expansion-related complications such as skin thinning, telangiectasia, and striae may result in expansion failure and ultimately jeopardize final outcome. In the past years, discontinuation of the expansion procedure was the only therapeutic option, when early alarm signs such as semitransparent appearance and telangiectasia of the expanded skin were encountered. We aimed to overcome these complications by therapeutic fat grafting to prevent skin necrosis and enable continuation of the expansion procedure.

Patients undergoing soft tissue expansion treatment for resurfacing skin lesions including scars and nevi that required therapeutic intervention due to early complication signs were included in this study. Patients were randomly divided into treatment group using autologous fat grafting and control group with discontinued expansion and expectant management. The treatment group received autologous fat transfer to the expanded skin.

ELIGIBILITY:
Inclusion Criteria:

* Expanding skin donor site at the face, neck, anterior chest wall, abdominal wall or back;
* Implanted silicone expander of 50 to 800 ml in size;
* History of deterioration in the expanded skin texture that did not improve after the inflation procedure was suspended for more than 2 weeks;
* Persistent high level of expander internal pressure;
* Need for further skin expansion;

Exclusion Criteria:

* Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for expansion; or history of delayed healing, radiational therapy;
* Rupture of expanded skin, expander exposure;
* Significant renal, cardiovascular, hepatic and psychiatric diseases;
* Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV);
* BMI less than 17 or insufficient subcutaneous fat;
* History of any hematological disease, including leukopenia , thrombocytopenia, or thrombocytosis;
* History of allogenic bone marrow transplantation;
* Pregnant or lactating woman;
* Long history of smoking;
* Evidence of malignant diseases or unwillingness to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To Measure the Change in Expansion Volume | Change from baseline volume at 12 weeks
  Record the volume(ml) of each expander
To Measure the Change in Skin Thickness | Change from baseline skin thickness at 12 weeks
  Record the thickness of the expanded skin(cm) by ultrasound scanning

SECONDARY OUTCOMES:
To Measure the Texture of Expanded Flap with VISIA scanner | baseline and 12 weeks post treatment
  Evaluate skin texture with VISIA scanner and compare the characteristics
Occurence of Major Adverse Events | Up to approximately 12 weeks after study start
  Including expanded flap ischaemia, necrosis, fluidify, infection, and all other adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China